CLINICAL TRIAL: NCT07346430
Title: Does Anxiety Affect Balance, Spasticity and Function in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor, Cairo University
Other Study IDs: P.T.REC/012/005784
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Anxiety; Spasticity
Keywords: anxiety; balance; spasticity; function; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Anxiety Disorders; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
children and adolescents with CP are at increased risk of developing mental health difficulties, particularly anxiety disorders, compared with their typically developing peers. this study was to investigate the correlation between anxiety, spasticity and balance in children with cerebral palsy.

DETAILED DESCRIPTION:
forty children with hemiplegia and diplegia were recruited from outpatient clinic of faculty of physical therapy, Cairo University and October 6 University. These children aged from 4 to 8 years old. Anxiety, motor function, spasticity and balance were assessed by Modified Yale Pre-Operative Anxiety Scale ((m -YPAS), The Gross Motor Functional Measurement-88 (GMFM-88), the modified Ashworth scale and Biodex balance system respectively.

ELIGIBILITY:
Inclusion Criteria:

* age 4-8 years from both genders
* diagnosed as hemiplegia and diplegia
* Gross Motor Function Classification System (GMFCS) levels I or II
* spasticity grade of 1 or I+ on the modified Ashworth Scale

Exclusion Criteria:

* significant visual, auditory, or perceptual deficits
* uncontrolled seizures
* acute illness

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: POWER statistical programming was used to test size estimation [Exact Correlation: Bivariate normal model, α = 0.05, β = 0.20, number of variables = 2, correlation ρH0 = 0, correlation ρH1 = 0.81, and coefficient of determination ρ2 = 0.66 and shown that the suitable sample size of current study was N = 13]. This coefficient of determination ρ2 was calculated from a pilot study of ten participants (between grades of spasticity and gross motor function).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
function | 3 months
  The Gross Motor Functional Measurement-88 used to measure function. The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item. SCORING KEY 0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes
spasticity | 3 months
  The modified Ashworth scale was used to measure spasticity. The test is performed by extending the patients limb's first from a position of maximal possible flexion to maximal possible extension (the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion.
  Scoring 0 No Increased in tone
  1. Slight increase in tone giving a catch when the limb is moved in flexion or extension 1+ Slight increase in muscle tone, indicated by a catch followed by minimal resistance throughout range of motion (ROM)
  2. More marked increase in tone through most of the ROM, but the limb easily flexed
  3. Considerable increase in tone, passive movement difficult
  4. Limb rigid in flexion or extension
balance | 3 months
  3. Biodex balance system was used to evaluate the postural stability and dynamic balance of children

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa s Ali, PhD, Principal Investigator — associate professor of physical therapy for pediatrics
Locations (1):
- Cairo University, Cairo, Egypt